CLINICAL TRIAL: NCT04216082
Title: A Single Center, Single-arm, Phase II Study of Anlotinib in Subjects With Advanced Malignancy
Brief Title: A Study of Anlotinib in Subjects With Advanced Malignancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-00-II
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Advanced Malignancy
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental): Anlotinib capsules given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib is a oral small molecule receptor tyrosine kinases inhibitor with the potency of inhibiting tumor angiogenesis as well as cell proliferation simultaneously and have been approved to treat advanced non-small cell lung cancer (NSCLC) in China. Anlotinib capsules given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).

SUMMARY:
Anlotinib is a tyrosine kinase inhibitors (TKI) with high effective in inhibiting angiogenesis and tumor cell proliferation by targeting VEGFR, PDGFR, FGFR and c-Kit. Previous phase I trial has shown the potency of anlotinib in treating patients with various cancer types who failed in standard treatment or lack proper treatment regimen. Here, a single center, single-arm, phase II study was conducted to further validate the efficacy and safety of anlotinib in these patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) 18~70 years old; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Life expectancy ≥ 3 months.

  2) Histopathologically confirmed advanced malignancy, including gynecological-related tumors, breast cancer, digestive tract tumors, melanoma, and gastrointestinal stromal tumors.

  3) Has no effective treatment choice, or failure/recurrence after conventional treatment.

  4) If has received chemotherapy, the treatment has been discontinued for at least 30 days.

  5) The main organs function are normally. 6) Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

  7) Understood and signed an informed consent form.

Exclusion Criteria:

* 1）Has other malignant tumors. 2) Has participated in other anticancer drug clinical trials within 4 weeks. 3) Has multiple factors affecting oral medication. 4) Has brain metastasis, spinal cord compression, cancerous meningitis. 5) Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1.

  6) Has any serious and / or uncontrolled disease. 7) Long-term unhealed wounds or fractures. 8) Has artery/venous thrombosis prior to the first dose within 6 months. 9) Has bleeding tendency or treated with anticoagulants or vitamin K antagonists.

  10) Has drug abuse history that unable to abstain from or mental disorders. 11)Has history of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation.

  12) According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2015-08-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Disease control rate（DCR） | up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 96 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China